CLINICAL TRIAL: NCT05356689
Title: Comparative Effects Of Patient Specific 3-Dimensional And 2-Dimensional Lumbar Traction On Pain And Functional Disability In Patients With Lumbar Radiculopathy
Brief Title: Patient Specific 3-Dimensional And 2-Dimensional Lumbar Traction In Patients With Lumbar Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0126 Hassan
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Lumbar Radiculopathy; Radiculopathy
Keywords: radiculopathy; lumber
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional physiotherapy (Experimental): Common Treatment: Hot pack (for 10 minutes), and US 1mhz for 7 minutes, Mackenzie exercises and cold pack will applied for 15 minutes after traction.
  Interventions: Other: mechanical traction
- 3- 2dimensional lumbar traction (Experimental): Group A: This group will get 3-dimensional lumbar traction on multi-dimensional traction bed spine MT. Group B: This group will get 2-dimensional lumbar traction on 2-dimensional traction bed.
  Interventions: Other: mechanical traction

INTERVENTIONS:
Other: mechanical traction — Group A: This group will get 3-dimensional lumbar traction on multi-dimensional traction bed spine MT. Group B: This group will get 2-dimensional lumbar traction on 2-dimensional traction bed. Common Treatment: Hot pack (for 10 minutes), and US 1mhz for 7 minutes, Mackenzie exercises and cold pack will applied for 15 minutes after traction.
  Other Names: core strengthening

SUMMARY:
The aim of study will be comparative effectiveness of the 2d and 3d lumbar traction on pain and functional disability in lumbar radiculopathy. This study will be useful for the physiotherapists to know which traction equipment will be more effective for the treatment of the lumbar radiculopathy

DETAILED DESCRIPTION:
In one studied the effect of patient-specific three-dimensional lumbar traction on pain and functional disability in individuals with lumbar intervertebral disc prolapse. Twenty-five participants (age range: 34-67 years) diagnosed with lumbar intervertebral disc prolapse were included in this study. Patient-specific three-dimensional lumbar traction was given as three sessions per week for the duration of one month. All participants completed a 10-cm visual analog pain scale and pain pressure threshold to assess pain and the Oswestry disability index to assess the functional disability. Twelve sessions of patient-specific three-dimensional lumbar traction promoted a reduction in pain and improvement in functional disability among subjects with lumbar intervertebral disc prolapse.Another studied to evaluate the effectiveness of traction in improving low back pain, functional outcome, and disk morphology in patients with herniated intervertebral disks. They included randomized control trials which involved adult patients with low back pain associated with herniated disk confirmed by magnetic resonance imaging or computed tomography, compared lumbar traction to sham or no traction, and provided quantitative measurements of pain and function before and after intervention. Methodological quality was assessed using the physiotherapy evidence database (Pedro) scale and Cochrane risk of bias assessment. Compared with sham or no traction, lumbar traction exhibited significantly more pain reduction and functional improvements in the short term, but not in the long term.

In Pakistan most of the physiotherapists used the two-dimensional traction bed for lumbar traction. There is insufficient study on Three-dimensional Traction unit. And there is no literature review is available on comparison of the 2d and 3d traction. To the best of researcher's knowledge, it can be concluded that insufficient literature is available on th

ELIGIBILITY:
Inclusion Criteria:

* Both male & female participants

  * Age group between 30 to 65 yrs.
  * Participants having chronic radiating pain in one or both legs will be included.
  * Patients having history of low back ache for 30 days in last six months.
  * Minimum of 25 score out of 100, on low back pain index
  * Participants suffering from intervertebral disc prolapse diagnosed by Orthopedic Surgeon or Experienced Physiotherapist

Exclusion Criteria:

* Participants having contraindication to spinal manipulative therapy. 18

  * Participants having disorders of autoimmune nature,
  * Participants having neurodegenerative diseases,
  * Participants having organic referred pain,
  * Participants having pregnancy,
  * participant with history of back surgery
  * History of cancer /metastasis
  * participant having medications periodically
  * participant suffering from psychological conditions
  * participants with history of inflammatory joint disease arthritis

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 10 months
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain". NPRS have shown high test-retest reliability (r = 0.96 and 0.95, respectively)
Oswestry Disability Index (ODI) | 10 months
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools The final score/index ranges from 0-100.
  A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound

CONTACTS AND LOCATIONS:
Overall Officials: saba Rafique, ppdpt, Principal Investigator — Riphah International University
Locations (1):
- Life Line Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tarulli AW, Raynor EM. Lumbosacral radiculopathy. Neurol Clin. 2007 May;25(2):387-405. doi: 10.1016/j.ncl.2007.01.008. PMID 17445735
- [Background] Schoenfeld AJ, Laughlin M, Bader JO, Bono CM. Characterization of the incidence and risk factors for the development of lumbar radiculopathy. J Spinal Disord Tech. 2012 May;25(3):163-7. doi: 10.1097/BSD.0b013e3182146e55. PMID 22543563
- [Background] Berry JA, Elia C, Saini HS, Miulli DE. A Review of Lumbar Radiculopathy, Diagnosis, and Treatment. Cureus. 2019 Oct 17;11(10):e5934. doi: 10.7759/cureus.5934. PMID 31788391
- [Background] Cheng YH, Hsu CY, Lin YN. The effect of mechanical traction on low back pain in patients with herniated intervertebral disks: a systemic review and meta-analysis. Clin Rehabil. 2020 Jan;34(1):13-22. doi: 10.1177/0269215519872528. Epub 2019 Aug 28. PMID 31456418